CLINICAL TRIAL: NCT02623244
Title: The Association Between Ovarian Endometrioma and Lower Urinary Tract Symptoms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Ob/Gyn, Far Eastern Memorial Hospital
Other Study IDs: 104120-F
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Endometrioma
Keywords: ovarian endometrioma; lower urinary tract symptoms; sexual dysfunction; gastrointestinal symptoms
MeSH Terms: conditions — Endometriosis; Lower Urinary Tract Symptoms; Sexual Dysfunction, Physiological | interventions — Ovariectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ovarian endometrioma: Women with ovarian endometrioma noted by ultrasonography.
  Interventions: Procedure: Laparoscopic oophorocystectomy or oophorectomy
- The control group: Women with age and body mass index matched and without ovarian endometrioma in ultrasonography

INTERVENTIONS:
Procedure: Laparoscopic oophorocystectomy or oophorectomy
  Groups: ovarian endometrioma

SUMMARY:
To assess the relationship between ovarian endometrioma and lower urinary tract symptoms, sexual function and gastrointestinal symptoms. In addition, the investigators also assess the impact of surgeries for ovarian endometrioma on lower urinary tract symptoms, sexual function and gastrointestinal symptoms.

DETAILED DESCRIPTION:
All patients were found to have ovarian endometrioma were invited to participate in this study. The size and location of ovarian endometrioma should be assessed by ultrasonography. Besides, all enrolled female patients will be asked to complete overactive bladder symptom score, female bladder function, female sexual function, and bowel incontinence assessment questionnaires and CA125 level. In addition, patients who underwent surgeries for ovarian endometrioma will be requested to complete the above questionnaires and CA125 check-up at 3 & 6 months after surgery. At least 30 women with age and body mass index matched and without ovarian endometrioma will be invited to participate in this study as the control group.

ELIGIBILITY:
Inclusion Criteria:

1. >20 years old.
2. Ovarian endometrioma: women having a frosted glass content in ovarian cyst

Exclusion Criteria:

1. The patient is acute lower urinary tract infection or intestinal inflammation.
2. Had received surgery bladder or urethra.
3. Patients with a history of urinary tract stones or tumors.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with ovarian endometrioma
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-11-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The association of ovarian endometrioma and overactive bladder symptoms score | 1 week
  The Spearman correlation between the presence of ovarian endometrioma and overactive bladder symptoms score

SECONDARY OUTCOMES:
The association between ovarian endometrioma and female sexual function index score | 1 weeks
  The Spearman correlation between the presence of ovarian endometrioma and female sexual function index score
The association between ovarian endometrioma and bowel incontinence assessment score | 1 weeks
  The Spearman correlation between the presence of ovarian endometrioma and bowel incontinence assessment score

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Mou Hsiao, MD, Principal Investigator — Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital, Banqiao, New Taipei, Taiwan
Locations (1):
- Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan